CLINICAL TRIAL: NCT04058158
Title: A Phase III Randomised, Double-blind, Multicentre Study to Compare the Efficacy, Safety, Pharmacokinetics, and Immunogenicity Between SB12 (Proposed Eculizumab Biosimilar) and Soliris® in Subjects With Paroxysmal Nocturnal Haemoglobinuria
Brief Title: A Study to Compare SB12 (Proposed Eculizumab Biosimilar) to Soliris in Subjects With Paroxysmal Nocturnal Haemoglobinuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB12-3003
Record Dates: First submitted 2019-08-12; First posted 2019-08-15 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — zwittergent 3-12; eculizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence I (Experimental): Subjects who are randomised to initially receive SB12 will be switched to receive Soliris® at Week 26
  Interventions: Drug: SB12 (proposed eculizumab biosimilar); Drug: Soliris (eculizumab)
- Treatment Sequence II (Experimental): Subjects who are randomised to initially receive Soliris® will be switched to receive SB12 at Week 26
  Interventions: Drug: SB12 (proposed eculizumab biosimilar); Drug: Soliris (eculizumab)

INTERVENTIONS:
Drug: SB12 (proposed eculizumab biosimilar) — 600 mg IV every week for first 4 weeks and 900 mg for the fifth week, followed by 900 mg every 2 weeks thereafter
Drug: Soliris (eculizumab) — 600 mg IV every week for first 4 weeks and 900 mg for the fifth week, followed by 900 mg every 2 weeks thereafter

SUMMARY:
This is a randomised Phase III, double-blind, multicentre, cross-over study to compare the efficacy, safety, pharmacokinetics, and immunogenicity between SB12 and Soliris® in subjects with PNH.

DETAILED DESCRIPTION:
Subjects will be randomised in a 1:1 ratio to either treatment sequence. Subjects randomly assigned to treatment with SB12 or Soliris® will receive 600 mg of eculizumab IV every week for first 4 weeks (initial phase) and 900 mg for the fifth week, followed by 900 mg every 2 weeks until Week 52. Subjects who are randomised to initially receive SB12 will be switched to receive Soliris® and subjects who are randomised to initially receive Soliris® will be switched to receive SB12 at Week 26.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or older
* Eculizumab-naïve patients with PNH
* Presence of the PNH white blood cell (WBC) clone ≥ 10%
* Documented LDH level ≥ 1.5 x ULN at Screening
* History of transfusion for anaemia within 12 months prior to Screening or having PNH-related symptoms at Screening
* Subjects must be vaccinated against Neisseria meningitides

Exclusion Criteria:

* Previous treatment with any complement pathway inhibitors
* ANC ≤ 500/mm3 or Platelet count < 70,000/mm3
* History of meningococcal disease
* History of bone marrow transplantation
* Known or suspected active bacterial/viral/fungal infection within 30 days
* Stable use of erythropoietic, corticosteroids, heparin, warfarin before randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-10-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- India (5):
  - Fortis Memorial Research Institute, Gurgaon, Haryana
  - Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh
  - Apollo Hospitals International Limited, Chennai
  - Amrita Institute of Medical Sciences and Research Centre, Kochi
  - Nil Ratan Sircar Medical College and Hospital, Kolkata
- Malaysia (5):
  - Hospital Ampang, Ampang
  - Hospital Sultanah Aminah, Johor Bahru
  - Queen Elizabeth Hospital - Kota Kinabalu, Kota Kinabalu
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Pulau Pinang, Pulau Pinang
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Tlalpan, Mexico
- Romania (4):
  - Colentina Clinical Hospital, Bucharest
  - Emergency University Hospital, Bucharest
  - Prof Dr I Chiricuta Institute of Oncology, Cluj-Napoca
  - Filantropia Municipal Clinical Hospital, Craiova
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Thailand (2):
  - Chulalongkorn University, Bangkok
  - Srinagarind Hospital, Nai Muang
- Ukraine (4):
  - Vinnytsia Regional Clinical Hospital n.a. M.I.Pyrohov, Vinnytsia, Vinnytsia Oblast
  - Municipal Institution Cherkasy Regional Oncology Dispensary of Cherkasy Regional Council, Cherkasy
  - Communal Non-profit Enterprise Regional Center of Oncology, Kharkiv
  - Poltava Regional Clinical Hospital n.a. M.V. Sklifosovskyi, Poltava

RESULTS

PARTICIPANT FLOW:
Groups:
- Soliris to SB12: Subjects randomly assigned to treatment with Soliris received 600 mg of eculizumab intravenous (IV) infusion every week for first 4 weeks (initial phase) and 900 mg for the fifth week, followed by 900 mg every 2 weeks thereafter.
- SB12 to Soliris: Subjects randomly assigned to treatment with SB12 received 600 mg of eculizumab intravenous (IV) infusion every week for first 4 weeks (initial phase) and 900 mg for the fifth week, followed by 900 mg every 2 weeks thereafter.
Period: Period 1
Arm/Group | Soliris to SB12 | SB12 to Soliris
Started | 25 | 25
Completed | 23 | 23
Not Completed | 2 | 2
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Pregnancy | 0 | 1
Period: Period 2
Arm/Group | Soliris to SB12 | SB12 to Soliris
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Soliris to SB12: Subjects randomly assigned to treatment with Soliris received 600 mg of eculizumab intravenous (IV) infusion every week for first 4 weeks (initial phase) and 900 mg for the fifth week, followed by 900 mg every 2 weeks thereafter. Subjects who were randomized to initially receive Soliris were switched to receive SB12 at Week 26.
- SB12 to Soliris: Subjects randomly assigned to treatment with SB12 received 600 mg of eculizumab intravenous (IV) infusion every week for first 4 weeks (initial phase) and 900 mg for the fifth week, followed by 900 mg every 2 weeks thereafter. Subjects who were randomized to initially receive SB12 were switched to receive Soliris at Week 26.
- Total: Total of all reporting groups
Arm/Group | Soliris to SB12 | SB12 to Soliris | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (13.67) | 40.0 (13.44) | 38.1 (13.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 11 | 17 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 15 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 7 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Lactate Dehydrogenase (U/L) at Week 26
Time Frame: Week 26
Population: Per-Protocol Set for LDH at a Single Time Point
Measure: Least Squares Mean (Standard Deviation); unit: U/L
Groups:
- SB12: SB12 treated group
- Soliris: Soliris treated group
Arm/Group | SB12 | Soliris
Number analyzed (Participants) | 23 | 23
U/L | 284.20 (456.73) | 249.72 (103.67)
Statistical Analysis 1: Comparison: SB12 vs Soliris; Test type: Equivalence — Pre-defined equivalence margin was [-337.2 to 337.2]; Least squares mean difference = 34.48, 95% CI 2-sided [-47.66 to 116.62]

2. Primary Outcome: Time-adjusted AUEC of LDH From Week 14 to Week 26 and From Week 40 to Week 52
Time Frame: From Week 14 to Week 26 and from Week 40 to Week 52
Population: Per-Protocol Set for AUEC of LDH
Measure: Geometric Least Squares Mean (Standard Deviation); unit: U/L
Arm/Group | SB12 | Soliris
Number analyzed (Participants) | 38 | 38
U/L | 279.65 (325.37) | 258.73 (95.09)
Statistical Analysis 1: Comparison: SB12 vs Soliris; Test type: Equivalence — Pre-defined equivalence margin was [0.77 to 1.29]; Ratio of geometric least squares mean = 1.08, 90% CI 2-sided [0.95 to 1.23]

ADVERSE EVENTS:
Time Frame: From the time of signing the informed consent form until Week 58 (EOS Visit) or ET Visit
Arm/Group | SB12 | Soliris
All-Cause Mortality (participants affected / at risk) | 0/47 | 1/47
Serious Adverse Events (participants affected / at risk) | 3/47 | 2/47
Other Adverse Events (participants affected / at risk) | 18/47 | 11/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB12 (N=47) | Soliris (N=47)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infusion site hypersensitivity (General disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB12 (N=47) | Soliris (N=47)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 2 (2)
Corona virus infection (Infections and infestations) | 8 (8) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 2 (4) | 3 (5)
Haemoglobinuria (Renal and urinary disorders) | 8 (15) | 2 (2)
Hypertension (Vascular disorders) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT04058158/Prot_SAP_000.pdf